CLINICAL TRIAL: NCT06399445
Title: The Effects of Nondepolarizing Muscle Relaxants During General Anesthesia on Perioperative and Postoperative Bleeding in Pediatric and Adult Patients Undergoing Tonsillectomy
Brief Title: Measurement of Blood Loss in Adenotonsillectomy During General Anesthesia According to the Application of Nondepolarizing Muscle Relaxants
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital of Split (Other)
Responsible Party: Principal Investigator, Ines Petrović, Principal Investigator, University Hospital of Split
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 2181-147/01-06/LJ.Z.-24-02
Record Dates: First submitted 2024-04-30; First posted 2024-05-03 (Actual); Last update posted 2024-05-03 (Actual); Status verified 2024-04

CONDITIONS: Anesthesia; Neuromuscular Blockade; Intraoperative Bleeding; Intraoperative Blood Loss; Post Operative Hemorrhage; Anesthesia Complication
Keywords: Adenotonsillectomy; Tonsillectomy; Intraoperative blood loss; Rocuronium bromide
MeSH Terms: conditions — Blood Loss, Surgical; Postoperative Hemorrhage | interventions — Rocuronium; Pharmaceutical Preparations

STUDY DESIGN:
Intervention Model Description: factorial randomised controlled trial
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- recurrent adenotonsillitis in the age group of 3 to 7 years old, non-rocuronium group (Placebo Comparator): Anesthetic management: after entering the operating room, the children will be monitored (electrodes for ECG, blood pressure cuff and pulse oximeter). We will use gas mixture of O2/N20 50/50% and concentration of Sevoflurane set between 5% and 6 % with a dose of 6 L/min (1.0 -1.3 MAC) for 10 breaths, then we will set 4 % concentration of Sevoflurane. After loss of consciousness, intravenous line 22 G will be obtained and 0.9 % saline infuse with a dose of 4 ml/kg/hr, Fentanyl 1 mcg/kg iv. and Propofol 2 mg/kg. During stage III of anesthetic depth, we will perform orotracheal intubation.
  Interventions: Procedure: conventional cold tonsillectomy and curettage adenoidectomy
- recurrent adenotonsillitis in the age group of 3 to 7 years old, rocuronium group (Active Comparator): Anesthetic management: after entering the operating room, chlidren will be monitored (electrodes for ECG, blood pressure cuff and pulse oximeter). We will use gas mixture of O2/N20 50/50% and concentration of Sevoflurane set between 5% and 6 % with a dose of 6 L/min (1.0 -1.3 MAC) for 10 breaths. After loss of consciousness, we will turn off Sevoflurane, intravenous line 22 G will be obtained and 0.9 % saline infuse with a dose of 4 ml/kg/hr, 1 mcg/kg Fentanyl, 2.5 mg/kg Propofol and 0.6 mg/kg Rocuronium bromide (esmeron). After 2 min, orotracheal intubation will be performed.
  Interventions: Procedure: conventional cold tonsillectomy and curettage adenoidectomy; Drug: Rocuronium Bromide

INTERVENTIONS:
Procedure: conventional cold tonsillectomy and curettage adenoidectomy — After entering the operating room, the children will be monitored (electrodes for ECG, blood pressure cuff and pulse oximeter). We will use gas mixture of O2/N20 50/50% and concentration of Sevoflurane set between 5% and 6 % with a dose of 6 L/min (1.0 -1.3 MAC) for 10 breaths, then we will set 4 % concentration of Sevoflurane. After loss of consciousness, intravenous line 22 G will be obtained and 0.9 % saline infuse with a dose of 4 ml/kg/hr, Fentanyl 1 mcg/kg iv. and Propofol 2 mg/kg. During stage III of anesthetic depth, we will perform orotracheal intubation.
Drug: Rocuronium Bromide — After entering the operating room, chlidren will be monitored (electrodes for ECG, blood pressure cuff and pulse oximeter). We will use gas mixture of O2/N20 50/50% and concentration of Sevoflurane set between 5% and 6 % with a dose of 6 L/min (1.0 -1.3 MAC) for 10 breaths. After loss of consciousness, we will turn off Sevoflurane, intravenous line 22 G will be obtained and 0.9 % saline infuse with a dose of 4 ml/kg/hr, 1 mcg/kg Fentanyl, 2.5 mg/kg Propofol and 0.6 mg/kg Rocuronium bromide (esmeron). After 2 min, orotracheal intubation will be performed.
  Other Names: Drug
  Arms: recurrent adenotonsillitis in the age group of 3 to 7 years old, rocuronium group

SUMMARY:
Although tonsillectomy is one of the most commonly performed surgeries, a review of literature reveals no articles dealing with the study of intraoperative blood loss in tonsillectomy and adenotonsillectomy according to the use of nondepolarizing muscle relaxants. The primary aim of our trial will be to compare blood loss in the operating theatre and postoperatively in two groups of children having adenotonsillectomy. The trial numbers will be randomised in blocks.

DETAILED DESCRIPTION:
Local clinical ethical committee approval is obtained. Written and oral informed consents of patients and parents of 60 chilldren will be obtained and the study initiated. Only American Society of Anesthesiologists (ASA) class I and II patients between 3 and 7 years of age will be eligible. The indication for surgery will be recurrent tonsillar infection and obstructive sleep apnea.

Totally 60 children aged between 3 and 7 years schedule for adenotonsillectomy will be included in this clinical randomized trial. All patients will be subjected to conventional cold tonsillectomy and curettage adenoidectomy under general anesthesia by the same surgeon.

The children will be monitored (electrodes for ECG, blood pressure cuff and pulse oximeter), intravenous line 22 G inserted and 0.9% saline solution 4 ml/kg/h infused. This procedure will be marked as A0 and will represent the beginning of anesthesia. For the induction of anesthesia, the children will be block randomized into two groups, rocuronium group and non-rocuronium group, each including 30 subjects. The randomisation list will be obtained from R program. In non-rocuronium group, we will perform inhalation induction with sevoflurane for tracheal intubation. In rocuronium group, 1 mcg/kg Fentanyl, 2.5 mg/kg Propofol and 0.6 mg/kg rocuronium bromide (esmeron) will be used for the induction of anesthesia. After 2 min, orotracheal intubation will be performed. Volume-controlled ventilation with a tidal volume of 7 ml/kg and a respiratory frequency of 14/min will be initiated in both groups. Every 5 minutes systolic, diastolic and mean arterial pressure(MAP) will be noticed along with heart rate and oxygen saturation by pulse oximetry(SpO2).

For the maintenance of anesthesia, we will use sevoflurane in 02/N20 mixture 50/50 %. Gas flow will continued until the end of the operation. In rocuronium group at the end of surgery, the neuromuscular blockade will be antagonized with Sugammadex 4 mg/kg, and extubation will be performed.

The time at with operator places the Boyle-Dawies mouth opener will mark start of the operation. The mentioned procedure will be marked as T0.

The time after detachment of the second tonsil will be designated as T1 and will indicate a point when hemostasis begins. Removal of the Boyle-Dawies opener and will be marked as T2.

Before starting the surgery, a good amount of cotton and ribbon gauze will be taken, weighed and sterilized. The suction bottle including the rubber tube will be cleaned and emptied completely before starting the operation. A known quantity of saline (100 ml) will be taken in the bowl and used for intermittent suction to prevent blockage of the suction tube.

During surgery, all the blood lost will be collected in the suction bottle. After adenoidectomy, a length of measured ribbon gauze piece (which will be taken from the measured pad) will be packed in the nasopharynx and left in position. Tonsillectomy will be then performed by dissecting the tonsil from the superior to inferior pole.The tonsillar fauces will be packed with cotton from the measured pad. Sterile surgical gauze, which are used for hemostasis within the operative area, will be weighed using an analytical balance before and after use. The resulting difference will represent the mass of lost blood in gauze and swabs. After ligating the bleeders, the nostrils and nasopharynx will be sucked. Then all the saline taken in the bowl will be sucked into the suction bottle. The suction tube will be raised above the level of the suction bottle to ensure that all the fluid was emptied into the suction bottle.

The sum of the above factors will represent the estimated blood loss in milliliters during adenotonsillectomy.

Postoperative hemoglobin and hematocrit will also be measured. Blood loss will be calculated by taking the average of actual blood loss and estimated blood loss

ELIGIBILITY:
Inclusion Criteria:

* conventional cold tonsillectomy and curettage adenoidectomy
* American Society of Anesthesiologists (ASA) physical status classification system: I, II aged between 3 and 7 years

Exclusion Criteria:

* Contraindications for general anesthesia, coagulation disorders, anemia,identification of an infection during systemic examinations

Ages: 3 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2024-04-18 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Intraoperative blood loss in milliliters | during surgery
  measurement of blood loss by the gravimetric method (the difference in the mass of surgical gauzes weighed on an analytical scale before and after hemostasis represents the mass of blood lost in the gauzes and swabs; we will convert the obtained number into milliliters by dividing it by 1,055 - specific blood density) , plus the volume of blood in the suction tank
Duration of hemostasis | during surgery
  Once the tonsils are snared off, we will measured time required to achieve hemostasis
Incidence of primary and secondary postoperative bleeding | up to 15 days after surgery
  Bleeding episodes are classified into primary hemorrhage within the first 24 hours of surgery and secondary hemorrhage after the first 24 hours of surgery. Our study will evaluate incidence of primary and secondary bleeding .

SECONDARY OUTCOMES:
Incidence of operative hemostasis due to postoperative primary and/or secondary hemorrhage | up to 15 days after surgery
  Incidence of postoperative hemorrhage requiring surgical treatment in general anesthesia
The number of consumed gauze and swabs in the rocuronium and non-rocuronium group | during surgery
  To evaluate number of the cotton balls soaked with blood in rocuronium and non-rocuronium group
Arterial blood pressure | during surgery
  Systolic, diastolic and mean arterial blood pressure changes every 5 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Ines Petrović, Principal Investigator — University Hospital Split, Department of Anesthesiology and Intensive Care, Split, Croatia; Ivan Vukovic, Study Chair — University Hospital Split, Department of Anesthesiology and Intensive Care, Split, Croatia; Benjamin Benzon, Study Chair — University of Split School of Medicine, Split, Croatia
Locations (1):
- University Hospital Split, Split, Croatia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Urik M, Bartos M, Sikolova S, Jancikova J, Perceova K, Jarkovsky J, Klabusayova E, Stourac P, Jabandziev P. Risk Factors for Postoperative Bleeding after Adenoidectomy. Children (Basel). 2021 Mar 21;8(3):242. doi: 10.3390/children8030242. PMID 33801025
- [Background] Alatas N, San I, Cengiz M, Iynen I, Yetkin A, Korkmaz B, Kar M. A mean red blood cell volume loss in tonsillectomy, adenoidectomy and adenotonsillectomy. Int J Pediatr Otorhinolaryngol. 2006 May;70(5):835-41. doi: 10.1016/j.ijporl.2005.09.011. Epub 2005 Oct 21. PMID 16243402
- [Background] Prasad KC, Prasad SC. Assessment of Operative Blood Loss and the Factors Affecting it in Tonsillectomy and Adenotonsillectomy. Indian J Otolaryngol Head Neck Surg. 2011 Oct;63(4):343-8. doi: 10.1007/s12070-011-0268-9. Epub 2011 Jun 3. PMID 23024939
- [Background] Apuhan T, Yildirim YS, Aksoy F, Borcin O, Ozturan O. The effects of desflurane and sevoflurane on the peri- and postoperative bleeding of adenotonsillectomy patients. Int J Pediatr Otorhinolaryngol. 2011 Jun;75(6):790-2. doi: 10.1016/j.ijporl.2011.03.008. Epub 2011 Apr 1. PMID 21458867
- [Background] Sarny S, Ossimitz G, Habermann W, Stammberger H. Hemorrhage following tonsil surgery: a multicenter prospective study. Laryngoscope. 2011 Dec;121(12):2553-60. doi: 10.1002/lary.22347. PMID 22109752